CLINICAL TRIAL: NCT01310595
Title: To Investigate the Effectiveness of Manual Therapy on Head-repositioning Accuracy and Static Postural Balance in Patients With Non-traumatic Chronic Mechanical Neck Pain.
Brief Title: Manual Therapy on Head-repositioning Accuracy and Static Postural Balance in Neck Pain Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Eddy Siu Hon Kit, Physiotherapist, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongKong PU
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Neck Pain
Keywords: Musculoskeletal manipulations; Proprioception; Postural balance
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual mobilization on cervical spine (Experimental): Manual mobilization given on cervical spine with infra-red therapy and self exercise and advice pamphlet.
  Interventions: Procedure: Manual mobilization on cervical spine
- Infra-red radiation therapy (Active Comparator): Infra-red radiation therapy with self exercise pamphlet given to patients with chronic mechanical neck pain.
  Interventions: Procedure: Infra-red therapy with self exercise pamphlet

INTERVENTIONS:
Procedure: Manual mobilization on cervical spine — Manual mobilization provided on selected cervical spine in patients with chronic mechanical neck apin
  Arms: Manual mobilization on cervical spine
Procedure: Infra-red therapy with self exercise pamphlet — Infra-red radiation therapy on cervical spine with self exercise pamphlet given to patients with chronic mechanical neck pain.
  Arms: Infra-red radiation therapy

SUMMARY:
To investigate the effect of cervical manual mobilization on head repositioning accuracy and postural balance in patients with chronic mechanical neck pain in a randomized controlled trial. Hypothesis: There is no difference between the intervention group (manual mobilization) and control group head repositioning accuracy and postural balance.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effectiveness of manual therapy to standing balance and head-neck proprioception sense in patients with chronic neck pain. The study will recruit 120 chronic neck pain patients and randomize the into 2 groups of 60. Group 1 will receive a course of manual therapy and infrared radiation for 15 minutes (twice weekly for 12 sessions). The other group (control) will receive infrared radiation therapy only. Manual therapy will be provided by experienced physiotherapists and assessed by a separate assessor. All outcome measures will be assessed at the beginning of study, upon completion of intervention, 3-month and 6-month after the completion of study. All measurements collected will be analysed by computerized statistical software in order to calculate the effectiveness of manual therapy and relationship among those outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Presented with a complaint of neck pain (defined as pain in the region from the upper thoracic spine to the occiput and the surrounding musculature) for more than 7 weeks.
* Had not received neck pain treatment in the past 1 month

Exclusion Criteria:

* Onset of presenting neck pain episode after trauma (eg, whiplash)
* History of cervical injury of trauma since the onset of presenting neck pain episode
* History of cervical injury or trauma
* Neck pain due to fracture, tumor, infection, severe spondyloarthropathy, or other non-mechanical cause such as inflammatory arthritis;
* Progressive neurological deficit, myelopathy, herniated nucleus pulpous, or severe incapacitating pain;
* Being treated by electrical devices;
* Blood coagulation disorder or were using corticosteroids or anticoagulant medications;
* History of stroke or transient ischemic attacks;
* Vertebrobasilar artery insufficiency;
* Neurologic disease (eg, multiple sclerosis, Parkinson's disease, syringomyelia);
* Congenital anomalies involving the C-spine;
* Systemic disease (eg, diabetes mellitus);
* Pain involving third-party liability or Workers' Compensation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Head repositioning accuracy | up to 6 month post intervention
  Head re-positioning accuracy by using laser-pointer mounted in a cyclist helmet.

SECONDARY OUTCOMES:
Postural balance | up to 6 month post intervention
  Standing postural sway using computerized validated equipment.
Northwick Park Questionnaire | up to 6 month post intervention
  Neck disability questionnaire
Active neck range of motion | up to 6 month post intervention
  Active neck range of motion using 3-dimensional goniometer.
Numeric Pain Rating Scale | up to 6 month post intervention
  Subjective numeric pain rating scale from 0 - 10.

CONTACTS AND LOCATIONS:
Overall Officials: Siu H Kit, MSc, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Physiotherapy Department, Prince of Wales Hospital, Stain, Hong Kong